CLINICAL TRIAL: NCT02466490
Title: A 24-week Trial of the Effectiveness and Safety of Fimasartan 60 mg Alone as Initial Treatment and Its Randomized Escalation to Fimasartan 120 mg or Fimasartan 60 mg/HCTZ 12.5 mg in Mexican Patients With Grade 1 and 2 Essential Hypertension
Brief Title: Efficacy and Safety of Fimasartan Alone or Combined With HCTZ in Mexican Patients With Essential Hypertension
Acronym: FIRME-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stendhal Americas, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIMA-MEX-12-01
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Hypertension, Essential
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fimasartan 60 mg Tablets (Experimental): FMS 60 mg tablets once a day during the initial 8 treatment weeks of the study
  Interventions: Drug: Fimasartan
- Fimasartan 120 mg Tablets (Active Comparator): FMS 120 mg tablets once a day during 4 weeks (treatment weeks 8 to 12)
  Interventions: Drug: Fimasartan
- Fimasartan; Hydrochlorothiazide 60/12.5 (Active Comparator): FMS 60 mg + HCTZ 12.5 mg tablets (fixed dose combination) once a day during 4 weeks (treatment weeks 8 to 12)
  Interventions: Drug: Fimasartan; Hydrochlorothiazide
- Fimasartan; Hydrochlorothiazide 120/12.5 (Experimental): FMS 120 mg + HCTZ 12.5 mg tablets (fixed dose combination) once a day during 12 weeks (treatment weeks 12 to 24)
  Interventions: Drug: Fimasartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: Fimasartan — Fimasartan tablets
  Other Names: Arakhor; Kanarb
  Arms: Fimasartan 120 mg Tablets; Fimasartan 60 mg Tablets
Drug: Fimasartan; Hydrochlorothiazide — Fimasartan plus hydrochlorothiazide fixed dose combination tablets
  Other Names: Diarakhor; Kanarb plus
  Arms: Fimasartan; Hydrochlorothiazide 120/12.5; Fimasartan; Hydrochlorothiazide 60/12.5

SUMMARY:
Fimasartan (FMS) is an AT1 receptor antagonist indicated for once a day administration, currently approved for the treatment of essential hypertension in Corea and Mexico. As the safety and efficacy of FMS was initially demonstrated in Korea only, it was necessary to address the potential for ethnic factors to have an effect on the drug´s efficacy and safety in the Mexican population. To address this need, a cohort of 272 Mexican subjects with grades 1-2 essential hypertension were sequentially treated on a treat to target basis (target: sitting Diastolic Blood Pressure (sDBP) <90 mmHg) with 60 mg FMS once a day (8 weeks), either 120 mg FMS or 60 mg FMS+12.5 mg HCTZ once a day (randomized 4 week treatment period) and 120 mg FMS once a day (during 12 weeks) for a total treatment period of 24 weeks.

DETAILED DESCRIPTION:
This was a prospective, open, multicentre, 24 week study of subjects with grade 1-2 essential hypertension eligible, according to the participating investigator's clinical judgement, to initial monotherapy.

Consenting, eligible subjects at 13 Mexican participating centers were initially assigned to monotherapy with 60 mg FMS once a day. At treatment week 8, those subjects with a sDBP ≥90 mmHg were randomized to either 120 mg FMS or to 60 mg FMS + 12.5 mg hydrochlorothiazide (HCTZ) once a day during 4 weeks. At treatment week 12, all non-responding subjects were finally assigned to 120 mg FMS + 12.5 mg HCTZ for the remaining 12 weeks of the planned 24 week treatment period. At treatment weeks 8 and 12, those subjects with a sDBP < 90 mmHg remained on their assigned treatment for the rest of the study.

This cohort study was designed to collect information on treatment effect (blood pressure changes from baseline/reference time and treatment response rates), and safety (i.e., incidence and characterization of clinical, laboratory and ECG adverse events); accordingly, subjects were assessed at treatment weeks 4, 8, 12, 16, 20 and 24 in terms of vital signs, clinical laboratory safety parameters, concomitant medications and adverse events. 12-lead ECG recordings were obtained from all subjects both at screening and at treatment week 24 and a subset of 11 subjects underwent both baseline and treatment week 8 24-hour ABPM recordings.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the study subject information and to voluntarily grant their informed consent.
* Men or women, 18 to 70 years old.
* With grade 1 or 2 essential arterial hypertension based on a sitting diastolic blood pressure (DBP) ≥90 mmHg and ≤109 mmHg (MEXICAN OFFICIAL NORM 030-SSA).
* Trustworthiness and willingness to attend all the study follow-up visits , according to the investigator's judgment.
* Patients already on antihypertensive therapy, not adequately controlled and that, according to the investigator's judgment, could be safely submitted to a two-week washout period.

Exclusion Criteria:

* Severe hypertension (Grade 3), with SBP≥180 mmHg and/or DBP≥110 mmHg, according to OFFICIAL MEXICAN NORM NOM 030-SSA criteria.
* Secondary hypertension.
* Impossibility to safely undergo a two week washout period from previous treatment prior to assignment to the study treatment, if applicable and according to the principal investigator´s judgment.
* Systemic diseases such as renal dysfunction (creatinine ≥1.5 time above the upper limit of the reference range), gastrointestinal disorders, hematological disorders or liver dysfunction (AST y/o ALT ≥1.5 times the upper limit of the reference range), capable to affect the absorption, distribution, metabolism and excretion of the study drug.
* Non-controlled diabetes mellitus (HbA1c>9%)
* Morbid obesity (BMI≥40 kg/m2)
* Myocardial infarction or severe coronary artery disease or clinically significant congestive heart failure, within the six months prior to the screening visit.
* Auto-immune or connective tissue disease.
* Evidence in the medical record of serious infectious diseases such as hepatitis type B or C or a positive HIV test at screening.
* Clinically significant laboratory test abnormalities, according to the investigator's judgment.
* Concomitant treatment which might affect blood pressure values.
* Known allergies or contraindication to the use of angiotensin II receptor antagonists.
* Pregnancy, breastfeeding or in the case of women with childbearing potential, the rejection to use an effective contraceptive method, according to the investigator's judgment.
* History of alcohol or addictive substance abuse.
* Subjects participating in other clinical studies or who have participated in other study within the 6 months prior to screening.
* Any other reason which in the investigator's opinion might contraindicate the participation of a subject in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Change From Baseline | Baseline to Treatment Week 8
  Treatment Week 8 mean sDBP and sitting Systolic Blood Pressure (SBP) changes from baseline (all study subjects treated with 60 mg FMS once a day)

SECONDARY OUTCOMES:
Blood Pressure Change from Week 8 | Treatment Week 8 to Treatment Week 12
  Treatment Week 12 mean sDBP and sSBP changes from week 8 on subjects randomized to either 120 mg FMS or 60 mg FMS + 12.5 mg HCTZ once a day
Week 8 Treatment Response Rate | Baseline to Treatment Week 8
  Proportion of subjects with sDBP < 90 mmHg at treatment week 8 (all subjects treated with 60 mg FMS once a day)
Week 12 Treatment Response Rate | Treatment Weeks 8 to 12
  Proportion of subjects with sDBP < 90 mmHg at treatment week 12 (subjects randomized to either 120 mg FMS or 60 mg FMS + 12.5 mg HCTZ once a day)
Blood Pressure Change from Week 12 | Treatment Weeks 12 to 24
  Treatment Week 24 mean sDBP and sSBP changes from treatment week 12 (subjects assigned at treatment week 12 to 120 mg FMS + 12.5 mg HCTZ
Week 24 Treatment Response Rate | Treatment Weeks 12 to 24
  Proportion of non-responding subjects assigned at treatment week 12 to 120 mg FMS + 12.5 mg HCTZ with sDBP < 90 mmHg at Treatment Week 24
Adverse Event Incidence | Baseline to Treatment Week 24
  Incidence and characterization of clinical, laboratory and ECG adverse events observed in all subjects assigned to treatment in the study receiving at least one dose of the study medications

OTHER OUTCOMES:
Pro-inflammatory marker changes from baseline | Baseline to treatment week 8
  Treatment Week 8 mean changes from baseline serum concentrations of hsCRP, adiponectin, ICAM-1 and IL6
Treatment Week 8 ABPM mean 24-hour BP changes from baseline | Baseline to treatment week 8
  Treatment week 8 mean 24-hour sDBP and sSBO changes from baseline in a subset of subjects with valid baseline and treatment week 8 ABPM recordings at two selected sites
Treatment Week 8 ABPM mean Daytime BP changes from baseline | Baseline to treatment week 8
  Treatment week 8 mean Daytime sDBP and sSBO changes from baseline in a subset of subjects with valid baseline and treatment week 8 ABPM recordings at two selected sites
Treatment Week 8 ABPM mean Nighttime BP changes from baseline | Baseline to treatment week 8
  Treatment week 8 mean Nighttime sDBP and sSBO changes from baseline in a subset of subjects with valid baseline and treatment week 8 ABPM recordings at two selected sites

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Conde-Carmona, M.D., Study Chair — Específicos Stendhal S.A. de C.V.
Locations (13):
- Mexico (13):
  - Hospital de Jesús IAP, México, D.f.
  - Hospital General de Ticomán, México, D.f.
  - Centro Médico Exel, Tijuana, Estado de Baja California
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Unidad de Investigación Clínica Cardiometabólica de Occidente, Guadalajara, Jalisco
  - Centro Universitario de Ciencias de la Salud, Universidad de Guadalajara, Guadalajara, Jalisco
  - Icle S.C., Guadalajara, Jalisco
  - Núcleo Médico La Paz, Guadalajara, Jalisco
  - Hospital Dr. Ángel Leaño, Zapopan, Jalisco
  - Instituto Jalisciense de Investigación en Diabetes y Obesidad S. C., Guadalajara, Jalsico
  - Cardiolink Clintrials, Monterrey, Nuevo León
  - Centro de Estudios Clínicos y Especialidades Médicas, Monterrey, Nuevo León
  - Hospital Dr. Ignacio Morones Prieto, San Luis Potosí City, San Luis Potosí

REFERENCES:
- [Result] Lee H, Yang HM, Lee HY, Kim JJ, Choi DJ, Seung KB, Jeon ES, Ha JW, Rim SJ, Park JB, Shin JH, Oh BH. Efficacy and tolerability of once-daily oral fimasartan 20 to 240 mg/d in Korean Patients with hypertension: findings from Two Phase II, randomized, double-blind, placebo-controlled studies. Clin Ther. 2012 Jun;34(6):1273-89. doi: 10.1016/j.clinthera.2012.04.021. Epub 2012 May 17. PMID 22608107
- [Result] Lee SE, Kim YJ, Lee HY, Yang HM, Park CG, Kim JJ, Kim SK, Rhee MY, Oh BH; Investigators. Efficacy and tolerability of fimasartan, a new angiotensin receptor blocker, compared with losartan (50/100 mg): a 12-week, phase III, multicenter, prospective, randomized, double-blind, parallel-group, dose escalation clinical trial with an optional 12-week extension phase in adult Korean patients with mild-to-moderate hypertension. Clin Ther. 2012 Mar;34(3):552-568, 568.e1-9. doi: 10.1016/j.clinthera.2012.01.024. Epub 2012 Mar 3. PMID 22381711
- [Result] Lee H, Kim KS, Chae SC, Jeong MH, Kim DS, Oh BH. Ambulatory blood pressure response to once-daily fimasartan: an 8-week, multicenter, randomized, double-blind, active-comparator, parallel-group study in Korean patients with mild to moderate essential hypertension. Clin Ther. 2013 Sep;35(9):1337-49. doi: 10.1016/j.clinthera.2013.06.021. Epub 2013 Aug 7. PMID 23932463
- [Result] Park JB, Sung KC, Kang SM, Cho EJ. Safety and efficacy of fimasartan in patients with arterial hypertension (Safe-KanArb study): an open-label observational study. Am J Cardiovasc Drugs. 2013 Feb;13(1):47-56. doi: 10.1007/s40256-013-0004-9. PMID 23344912
- [Result] Chi YH, Lee H, Paik SH, Lee JH, Yoo BW, Kim JH, Tan HK, Kim SL. Safety, tolerability, pharmacokinetics, and pharmacodynamics of fimasartan following single and repeated oral administration in the fasted and fed states in healthy subjects. Am J Cardiovasc Drugs. 2011 Oct 1;11(5):335-46. doi: 10.2165/11593840-000000000-00000. PMID 21910510
- [Result] Madamanchi NR, Vendrov A, Runge MS. Oxidative stress and vascular disease. Arterioscler Thromb Vasc Biol. 2005 Jan;25(1):29-38. doi: 10.1161/01.ATV.0000150649.39934.13. Epub 2004 Nov 11. PMID 15539615